CLINICAL TRIAL: NCT04931030
Title: Effects of Low Carbohydrate Diet (LCBD) on Weight and Renal Outcome in Patients With Diabetic Kidney Disease (DKD)- A Pilot Study
Brief Title: Low Carbohydrate Diet in Diabetic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Teknologi Mara (Other)
Collaborators: IMU University, Malaysia (Other)
Responsible Party: Principal Investigator, Rohana Abdul Ghani, Deputy Dean Postgraduate Studies and Professional Training, Principal Investigator, Clinical Professor in Medicine, Universiti Teknologi Mara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 600-IRMI (5/1/6)
Record Dates: First submitted 2021-06-01; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Type 2 Diabetes Mellitus; Diabetic Kidney Disease; Obesity
Keywords: low carbohydrate diet; chronic kidney disease; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies; Obesity; Renal Insufficiency, Chronic; Diabetes Mellitus | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, unblinded, dietary intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low carbohydrate diet (LCBD) (Experimental): Subjects are given a dietary prescription of 20g of carbohydrate daily in addition to standard low protein diet of 0.6-0.7g/kg/day and low salt diet.
  Interventions: Other: Dietary advice
- Low protein diet only (LPD) (No Intervention): Subjects are given the standard dietary advice of chronic kidney disease of low protein diet of 0.6-0.7g/kg/day and low salt diet.

INTERVENTIONS:
Other: Dietary advice — Subjects are provided dietary advice by the dietitians as part of the research team/ investigators
  Arms: Low carbohydrate diet (LCBD)

SUMMARY:
The current population of type 2 diabetes mellitus (T2DM) worldwide is over 200 million and Malaysia contributes to 1.2% of that number. The prevalence of T2DM in Malaysia has approximately tripled over the last three decades from 6.3% in 1986 to 17.5% of the adult population in 2015.T2DM is a progressive disease associated with debilitating microvascular and macrovascular complications. The prevalence of chronic kidney disease (CKD) in Peninsular Malaysia was high at 9.1% of the adult population in 2011. T2DM is the leading cause of renal failure for patients commencing dialysis, increasing from 53% of new dialysis patients in 2004 to 61% in 2013. Therefore, diabetic kidney disease (DKD) is a debilitating complication which not only imposes significant health problems but also confers financial burden on affected patients. There has been increasing amount of understanding in the complexity of the relationship between T2DM and obesity. As the prevalence of both conditions continue to demonstrate a parallel rise, the influence of obesity on T2DM is further marked. Thus, this has led to greater emphasis on weight loss in the management of T2DM. More recent anti-diabetic medications including SGLT-2 inhibitors and GLP1 agonists demonstrated greater efficacy in improving glycaemic control and their ability to produce weight reduction. In addition, there has been more interest in the effects of these drugs on retardation of renal disease progression. The mechanism is unclear, either attributed by direct drug effects on renal glomerular-tubular structures, through the Renin-Angiotensin-Aldosterone-System (RAAS), or other pathways. Another pausible explanation is the significant weight loss, which has been shown to have a significant effect of attenuation of renal disease.

Weight reduction programs have long been a complex and tedious treatment plan which has inconsistent, non-duplicable and unpredictable outcomes. Most programs emphasized on medical nutrition therapy and lifestyle changes. There has been many different dietary plans which share a common goal ie to reduce calori intake whilst increasing energy expenditure. Few have been successfully reproducible, limited by either patient adherence or modest outcome.

Low carbohydrate diet is a diet plan which stresses on reducing carbohydrate intake to less than 20g daily. Numerous studies have shown that weight loss could be obtained by reduction of calori intake in either the form of carbohydrate or fat. CKD patients are recommended to consume low protein diet of less than 0.6-0.7g/kg/day with little emphasis on calori or carbohydrate intake.

This study, thus, aims to evaluate the effects of low carbohydrate and moderate fat (LCBD) in addition to low protein diet on renal disease in patients with DKD.

DETAILED DESCRIPTION:
This is an investigator-initiated, single center, randomized, controlled, clinical trial in Type 2 diabetes mellitus patients, comparing 16-weeks of LCBD compared to standard medical therapy in patients with DKD.

Patients would be recruited from the Endocrinology and Nephrology clinics in UiTM Medical Specialist Center. Inclusion criteria would include patients aged between 40-75 years old, diagnosis with Type 2 DM of more than 5 years with stable CKD stage 2 and 3 of more than 6 months, HbA1c of 7% - 10.5%.

Exclusion Criteria include patients with Type 1 DM, experiencing frequent hypoglycaemia, abnormal liver function tests, heart failure (New York Heart Association functional class III-IV), active systemic inflammatory disease, chronic renal failure requiring hemodialysis, active hepatic disease and collagen disease, malignancy, recent hospital admission within the past 3 months, pregnant women, breastfeeding or planning to conceive within the next year.

Following informed consent, patients would be randomised to either LCBD or low protein Diet (LPD) group.

All recruited patients will be given the standard dietary and exercise advice which will include low protein of 0.6-0.7g/kg/day and low salt diet.

In addition, patients within the LCBD will be given a prescription diet of 20g of carbohydrate daily. This will be supplemented by visual aids on carbohydrate counts of various local food. Patients would be given the option to choose their most appropriate food types which will amount to the carbohydrate count given. Patients on oral anti-diabetic treatment including insulin will advised on titrations of their medications to avoid hypoglycaemia.

The control arm will not be given any additional advice. All patients will be required to fill in a 3-day food diary during their scheduled visits which will be at 8 weeks and 16 weeks.

Clinical assessments include blood sampling of approximately 8 ml which will be done at baseline and at study end.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosed with Type 2 DM of more than 5 years
2. Diagnosis of stable CKD of more than 6 months
3. CKD stage 2 and 3
4. HbA1c of 7% - 10.5%
5. Patient age between 40-75 years old
6. Able to sign informed consent

Exclusion Criteria

1. Type 1 DM
2. Frequent hypoglycaemia
3. Persistent elevations of serum transminase
4. Heart failure (New York Heart Association functional class III-IV), active systemic inflammatory disease, chronic renal failure requiring hemodialysis, active hepatic disease and collagen disease
5. Malignancy
6. Recent hospital admission for acute within the past 3 months
7. Pregnant women, breastfeeding or planning to conceive within the next year

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline serum Creatinine at 12 weeks | Study end at 12 weeks
  Creatinine in micromol/L
Change from baseline urine microalbuminuria at 12 weeks | Study end at 12 weeks
  Urine microalbuminuria in mmol/L

SECONDARY OUTCOMES:
Change from baseline HbA1c at 12 weeks | Study end at 12 weeks
  HbA1c in %
Change from baseline fasting plasma glucose at 12 weeks | Study end at 12 weeks
  FPG in mmol/L
Change from baseline lipid levels at 12 weeks | Study end at 12 weeks
  Cholesterol in mmol/L
Change from baseline weight at 12 weeks | Study end at 12 weeks
  Weight in kg
Change from baseline hip circumference (HC) at 12 weeks | Study end at 12 weeks
  HC in cm
Change from baseline waist circumference (WC) at 12 weeks | Study end at 12 weeks
  WC in cm
Change from baseline estimated visceral adispose tissue (Est VAT) at 12 weeks | Study end at 12 weeks
  Est VAT in %
Change from baseline blood pressure at 12 weeks | Study end at 12 weeks
  Blood pressure in mmHg
Change from baseline highly sensitivity C-reactive protein (hsCRP) at 12 weeks | Study end at 12 weeks
  hsCRP in nmol/L
Change from baseline Interleukin-6 (IL-6) at 12 weeks | Study end at 12 weeks
  IL-6 in pg/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Teknologi MARA, Petaling Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Unidentified subjects' raw data is required for some journal submissions

REFERENCES:
- [Background] Feisul MI, Azmi S. (Eds). National Diabetes Registry Report, Volume 1, 2009-2012. Kuala Lumpur; Ministry of Health Malaysia; 2013 Jul.
- [Background] National Health and Morbidity Survey 2015 (NHMS 2015). Ministry of Health, Kuala Lumpur, Malaysia
- [Background] Hooi LS, Ong LM, Ahmad G, Bavanandan S, Ahmad NA, Naidu BM, Mohamud WN, Yusoff MF. A population-based study measuring the prevalence of chronic kidney disease among adults in West Malaysia. Kidney Int. 2013 Nov;84(5):1034-40. doi: 10.1038/ki.2013.220. Epub 2013 Jun 12. PMID 23760287
- [Background] B. Goh, L. Ong, Y. Lim. Twenty First Report of the Malaysian Dialysis and Transplant 2013. Malaysian Society of Nephrology, Kuala Lumpur, Malaysia (2014)

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT04931030/Prot_SAP_ICF_000.pdf